CLINICAL TRIAL: NCT04406545
Title: Investigation of Systemic Microvascular Flow and Reactivity in Patients Presenting in the Acute Phase of Coronavirus Disease-19.
Brief Title: Microvascular Flow and Reactivity in Patients Presenting in the Acute Phase of COVID-19.
Status: Completed | Type: Observational
Sponsor: National Institute of Cardiology, Laranjeiras, Brazil (Other Government)
Responsible Party: Principal Investigator, Eduardo Tibirica, MD, PhD, Senior Researcher, National Institute of Cardiology, Laranjeiras, Brazil
Other Study IDs: #CAAE 31237220.1.0000.5272
Record Dates: First submitted 2020-05-23; First posted 2020-05-28 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Coronavirus Infection; Endothelial Dysfunction; Microvascular Rarefaction
MeSH Terms: conditions — Coronavirus Infections; Microvascular Rarefaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — ultra frozen plasma samples will be stocked for the evaluation of inflammatory anti-inflammatory cytokines
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- healthy volunteers: skin laser Doppler perfusion monitoring before and after local thermal hyperemia
  Interventions: Other: evaluation of skin microvascular flow and reactivity
- cardiovascular disease and COVID-19 infection: skin laser Doppler perfusion monitoring before and after local thermal hyperemia
  Interventions: Other: evaluation of skin microvascular flow and reactivity
- cardiovascular disease without COVID-19 infection: skin laser Doppler perfusion monitoring before and after local thermal hyperemia

INTERVENTIONS:
Other: evaluation of skin microvascular flow and reactivity — evaluation of skin microvascular flow and reactivity using laser Doppler perfusion monitoring
  Groups: cardiovascular disease and COVID-19 infection; healthy volunteers

SUMMARY:
Considering that the intensity of systemic microvascular changes in patients in the acute phase of COVID-19 could be related to disease progression and prognosis, the present cross-sectional and observational study aims to investigate the presence of endothelial dysfunction in these patients, also looking for to evaluate associations between the presence of endothelial dysfunction and demographic, clinical and laboratory variables.

DETAILED DESCRIPTION:
An association between the presence of previous cardiovascular disease and adverse prognosis has been demonstrated in patients with COVID-19 (coronavirus disease-19), presenting increases of up to 5-10 times in mortality.

As an initial process, the SARS-CoV-2 virus, anchored in the transmembrane angiotensin-converting enzyme 2 (ECA2), penetrates host cells, including endothelial cells, pericytes and macrophages, in addition to type II pneumocytes.

Cellular invasion results in massive release of several pro-inflammatory cytokines ("cytokine storm"), such as IL-1β, IFN-1 and IL-6, by the cells of the immune system. In turn, cytokines increase the process of vascular inflammation and the expression of leukocyte-vascular endothelium adhesion proteins, which results in endothelial activation accompanied by a pro-coagulant and pro-adhesive phenotype - between leukocytes, platelets, red blood cells and vascular endothelium - characteristic of the dysfunctional endothelium in the microcirculation, which results in severe changes in the microvascular flow and, as a result, in tissue perfusion.

It is also worth noting that the patients most vulnerable to the development of complications are those with pre-existing endothelial dysfunction, associated with several risk factors such as male gender and smoking, and comorbidities such as hypertension, diabetes and obesity, all of which are associated with poor prognosis in COVID -19.

Considering that the intensity of systemic microvascular changes in patients in the acute phase of COVID-19 could be related to disease progression and prognosis, the present cross-sectional and observational study aims to investigate the presence of endothelial dysfunction in these patients, also evaluating associations between the presence of endothelial dysfunction and demographic, clinical and laboratory variables.

ELIGIBILITY:
* Age> 18 years admitted to the hospital
* SARS-CoV-2 positive real-time PCR molecular test

Exclusion Criteria:

* Presence of non-COVID infection with systemic and microbiologically documented repercussions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: - We will include adult patients will with SARS-CoV-2 positive RT-PCR, admitted to the hospital in a ward or intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
To evaluate, through laser doppler, the presence of changes in systemic microvascular endothelial function in patients in the acute phase of COVID-19. | Microvascular reactivity will be evaluated after a 20-minute rest in the supine position in a temperature-controlled room.
  skin laser Doppler perfusion monitoring before and after local thermal hyperemia

SECONDARY OUTCOMES:
To evaluate, using laser Doppler perfusion monitoring, the presence of changes in systemic microvascular endothelial function in patients twelve months after COVID-19 recovery. | Microvascular reactivity will be evaluated after a 20-minute rest in the supine position in a temperature-controlled room
  Skin laser Doppler perfusion monitoring before and after local thermal hyperemia

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Cardiology, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided